CLINICAL TRIAL: NCT03339973
Title: A Randomised, Placebo-controlled, Double-blind, Interventional, Multicenter, Phase I/IIa Clinical Trial to Investigate the Efficacy and Safety of Allo-APZ2-PAOD for the Treatment of Peripheral Arterial Occlusive Disease (PAOD)
Brief Title: Allogeneic ABCB5-positive Stem Cells for Treatment of PAOD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Very slow recruitment of patients and the current COVID-19 pandemic situation.
Sponsor: RHEACELL GmbH & Co. KG (Industry)
Collaborators: FGK Clinical Research GmbH (Industry); Ticeba GmbH (Industry); Granzer Regulatory Consulting & Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: allo-APZ2-PAOD-II-01
Record Dates: First submitted 2017-10-11; First posted 2017-11-13 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Peripheral Arterial Occlusive Disease
Keywords: Peripheral Arterial Occlusive Disease; ABCB5; allogeneic; mesenchymal stem cells; advanced therapy medicinal product; somatic cell therapy; phase I/IIa; non-healing ulcers
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind, interventional, multicenter, phase I/IIa clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- allo-APZ2-PAOD (Experimental): 20-30 intramuscular injections, single dose of allo-APZ2-PAOD, 150 - 225 x 10^6 cells per patient (depending on length of lower leg)
  Interventions: Biological: allo-APZ2-PAOD
- Placebo (Placebo Comparator): 20-30 intramuscular injections, vehicle solution (depending on length of lower leg)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: allo-APZ2-PAOD — Suspension of ABCB5-positive mesenchymal stem cells in pre-filled syringe
  Arms: allo-APZ2-PAOD
Drug: Placebo — Solution for injection in pre-filled syringe
  Arms: Placebo

SUMMARY:
The aim of this clinical trial is to investigate the efficacy (by monitoring the wound size reduction of Peripheral Arterial Occlusive Disease-related clinically relevant ulcers) and safety (by monitoring adverse events) of one dose of allo-APZ2-PAOD administered intramuscularly into an affected lower leg of patients with Peripheral Arterial Occlusive Disease.

DETAILED DESCRIPTION:
This is an interventional, randomised, placebo-controlled, double-blind phase I/IIa clinical trial to investigate the efficacy and safety of allo-APZ2-PAOD for the treatment of Peripheral Arterial Occlusive Disease patients with non-healing ulcers. The allogeneic investigational product allo-APZ2-PAOD contains skin-derived ABCB5-positive mesenchymal stem cells isolated from skin tissue of healthy donors and stored in a donor cell bank.

Patients are followed up for efficacy for 12 weeks by clinical visits at the clinical trial sites to monitor wound healing. The wound healing process of all relevant ulcers will be documented by standardized photography and the quality of the wound healing process will be assessed.

Pain will be assessed using a numerical rating scale and quality of life will be investigated with a standardized and validated questionnaire. To assess long-term safety of allo-APZ2-PAOD three follow-up visits at Months 6, 9 and 12 post IMP applications are included. An unblinded external Independent Data Monitoring Committee (IDMC) will continuously monitor safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 45 to 85 years;
2. Patients having PAOD clinically confirmed (maximal systolic ankle pressures ≤ 70 mmHg or systolic toe pressures ≤ 50 mmHg or transcutaneous partial oxygen pressures (tcp02) ≤ 30 mmHg in supine position) as Rutherford category 5 in at least one lower extremity;
3. Angiography results (DSA, CTA or MRA) for the localization of the high-grade obstruction of an artery of the affected leg (≥ 70 %) that is the leading cause for the ulceration are present and not older than 3 months;
4. One or more clinically relevant and quantifiable ulcer(s) below the ankle with a minimum size of 0.5 cm² per ulcer and a maximum wound size of 20 cm² for all ulcers together;
5. Positive vote of the Advisory Board on the suitability of the wound(s) for enrolment, based on the wound photographs;
6. Patients not eligible for surgical/interventional reconstruction due to technical limitations or comorbidity;
7. No evidence of wound healing after standard of care treatment for at least 1 week before screening;
8. In Patients suffering from 2 or more ulcers at the same extremity, these ulcers must be separated by a minimum bridge of 1 cm of epithelialized skin;
9. If patients are hypertensive, they have to be treated with anti-hypertensive medication according to the applicable guideline;
10. Body mass index (BMI) between 20 and 40 kg/m²;
11. Women of childbearing potential must have a negative blood pregnancy test at screening;
12. Women of childbearing potential and their partner must be willing to use highly effective contraceptive methods during the course of the clinical trial;
13. Patients must be able to consent, have been informed of the nature, the scope and the relevance of the study, voluntarily agree to participation and the study's provisions, and have duly signed the ICF. Subject agrees to comply with the protocol-mandated procedures and visits.

Exclusion Criteria:

1. Patients with skin lesions of leading venous origin or patients suffering from a vasculitis;
2. Patients with thrombangiitis obliterans;
3. Diabetic patients in whom the leading cause for lesions is microangiopathy or neuropathy;
4. Patients with high grade obstruction (≥ 70 %) in the aorto-iliac segment or the common femoral artery as leading cause for skin lesions;
5. Patients with ulcers at the heel due to immobility;
6. Patients with osteomyelitis at ulceration;
7. Patients medicated with vitamin K antagonist, if treatment cannot be stopped before injection or bridged according to applicable guidelines;
8. Patients medicated with DOACs, if they cannot be withheld for 24 hours before injection;
9. Surgical/interventional reconstruction during 1 week before screening (not applicable if it becomes evident during reconstruction that revascularization is not successful: these patients can be included immediately);
10. Patients for whom major amputation is scheduled on target leg;
11. Patients with uncontrolled hypertension defined as systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg; For these patients a re-screening and inclusion into the study will be possible after blood pressure is controlled;
12. Patients who had a myocardial infarction during 3 months before screening;
13. Patients with uncontrolled infection at any of the relevant ulcers;
14. Patients with uncontrolled acute or chronic infection with systemic symptoms;
15. Known serious disease with life expectancy of less than 1 year;
16. Any chronic dermatological disorders diagnosed at the investigator's discretion;
17. Skin disorders, unrelated to the ulcer, that are present adjacent to any of the relevant ulcers;
18. Active malignancy or history of malignancy within 5 years prior to study entry;
19. Patients tested positive for human immunodeficiency virus (HIV˗1, HIV-2), Hepatitis B or Hepatitis C;
20. Any known allergies to components of the IMP;
21. Current or previous (within 30 days of enrolment) treatment with another IMP, or participation and/or under follow-up in another clinical trial;
22. Current use of glucocorticoid-medication above Cushing threshold dose (>7.5 mg/d prednisone or equivalent) or any other prohibited medication or therapy;
23. Known abuse of alcohol, drugs, or medicinal products;
24. Patients anticipated to be unwilling or unable to comply with the requirements of the protocol;
25. Evidence of any other medical conditions (such as psychiatric illness, physical examination, or laboratory findings) that may interfere with the planned treatment, affect the patient's compliance, or place the patient at high risk of complications related to the treatment;
26. Pregnant or lactating woman;
27. Employees of the sponsor, or employees or relatives of the investigator.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline to week 12 in total wound size of the target leg | Week 12, or last available post-baseline measurement if the Week 12 measurement is missing.
  Percent change from baseline to week 12 in total wound size of the target leg will be evaluated. The total wound size of the target leg is calculated as sum of the wound sizes of all relevant ulcers of the target leg.
Assessment of adverse event (AE) occurrence | Up to 12 months.
  All AEs occurring during the clinical trial will be registered, documented and evaluated.

SECONDARY OUTCOMES:
Time to total healing of all relevant ulcers at target leg | A priori specification not possible; between baseline and week 12 post baseline.
  Time to total healing of all relevant ulcers at target leg will be evaluated.
Percent change in total wound size of the target leg | Baseline, week 1, 2, 4, 6, and 8.
  Percent change in total wound size of the target leg will be evaluated.
Absolute change in total wound size of the target leg | Baseline, week 1, 2, 4, 6, 8 and 12.
  Absolute change in total wound size of the target leg will be evaluated.
Ankle-brachial index (ABI) of target leg; | Screening Visit, Baseline, Week 2, 4, 8 and 12.
  Ankle-brachial index (ABI) of target leg will be evaluated.
Number of amputated toes at target leg | A priori specification not possible; between baseline and week 12 post baseline.
  Number of amputated toes at target leg will be registered, documented and evaluated.
Time to major amputation at target leg until week 12; | A priori specification not possible; between baseline and week 12 post baseline.
  Time to major amputation at target leg until week 12 will be evaluated.
Assessment of epithelialization in % of wound area of all relevant ulcers of the target leg | Day 0 prior IMP-application, week 2, 4, 8 and 12.
  Epithelialization of all relevant ulcers of the target leg will be evaluated by the investigator based on image analysis for each ulcer individually.
Assessment of further wound healing parameters: formation of granulation tissue in % of wound area and wound exudation of all relevant ulcers of the target leg | Day 0 prior IMP-application, week 2, 4, 8 and 12.
  Formation of granulation tissue in % of wound area will be assessed by the investigator based on image analysis for each ulcer individually.
  Wound exudation of all relevant ulcers of the target leg will be evaluated as high-moderate-low based on amounts of fluid on the wound.
Assessment of quality of life (QoL) using the short form 36 (SF-36) questionnaire | Day 0 prior IMP-application, week 2, 8 and 12.
  Quality of life (QoL) using the short form 36 (SF-36) questionnaire will be evaluated.
  The SF-36 questionnaire is a self-administered questionnaire containing 36 items.
  It measures health on eight multi-item dimensions, covering functional status, well being, and overall evaluation of health.
Pain assessment as per numerical rating scale (NRS). | Day 0 prior IMP-application, week 2, 4, 8 and 12.
  Pain assessment as per numerical rating scale (NRS) will be evaluated.
Physical examination at week 12; | Week 12.
  A full physical examination will be performed at week 12 and abnormal physical examination results will be evaluated and reported as AEs.
Vital signs: Body temperature at week 12; | Week 12.
  Body temperature at week 12 will be evaluated.
Vital signs: Blood pressure at week 12; | Week 12.
  Blood pressure at week 12 will be evaluated.
Vital signs: Heart rate at week 12; | Week 12.
  Heart rate at week 12 will be evaluated.
Assessment of Laboratory values (Hematology) at Week 12: | Week 12.
  The Hematology values will be measured and evaluated at Week 12
Assessment of Laboratory values (Clinical chemistry) at Week 12 | Week 12.
  The clinical chemistry values will be measured and evaluated at Week 12.
Time to major amputation | A priori specification not possible; between baseline and month 12 post baseline.
  Time to major amputation will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Müller, Prof. Dr., Principal Investigator — Christian-Albrechts-Universität zu Kiel, Klinik für Innere Medizin III Kardiologie, Angiologie und internistische Intensivmedizin, Kiel, Germany
Locations (18):
- Austria (3):
  - LKH-Univ. Klinikum Graz, Graz
  - Konventhospital der Barmherzigen Brüder Linz, Linz
  - Hanusch-Krankenhaus Wien, Vienna
- Krajská zdravotní a.s. - Masarykova nemocnice v Ústí nad Labem, o.z., Ústí nad Labem, Czechia
- Germany (12):
  - Franziskus-Krankenhaus Berlin, Berlin
  - Universitätsklinikum "Carl Gustav Carus" der TU Dresden, Dresden
  - Helios Weißeritztal-Kliniken Klinikum Freital, Freital
  - Universitäres Herzzentrum Hamburg GmbH (UHZ), Hamburg
  - Asklepios Klinikum Harburg, Hamburg
  - St. Josefskrankenhaus Heidelberg GmbH, Heidelberg
  - Universitätsklinikum Heidelberg, Heidelberg
  - SRH Klinikum Karlsbad-Langensteinbach GmbH, Karlsbad
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Mannheim, Mannheim
  - Klinikum der Universität München, Campus Innenstadt, München
  - Medizinisches Versorgungszentrum der Barmherzigen Brüder Trier, Trier
- Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan, Poland
- East Surrey Hospital, Surrey and Sussex Healthcare NHS Trust, Redhill, United Kingdom

IPD SHARING:
Plan to Share IPD: No